CLINICAL TRIAL: NCT04950608
Title: Pilot Study of Psilocybin-Assisted Therapy for Demoralization in Patients Receiving Hospice Care - PATH Study
Brief Title: Pilot Study of Psilocybin-Assisted Therapy for Demoralization in Patients Receiving Hospice Care
Acronym: PATH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yvan Beaussant, MD, MSci (Other)
Collaborators: Oppenheimer Family Psychosocial Oncology and Palliative Care Research Grants (Unknown); Usona Institute (Other); Carey and Claudia Turnbull Family Foundation (Unknown); Heffter Research Institute (Other); George Sarlo Foundation (Unknown); RiverStyx Foundation (Other); Council on Spiritual Practices Fund at the San Francisco Foundation (Unknown); Nikean Foundation (Unknown); Jack Smith (Unknown)
Responsible Party: Sponsor-Investigator, Yvan Beaussant, MD, MSci, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-202
Record Dates: First submitted 2021-06-09; First posted 2021-07-06 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hospice; Psilocybin; Demoralization; Terminal Illness; Cancer-related Problem/Condition; Psychotherapy; Terminal Cancer; Cancer Terminal
Keywords: Hospice; Psilocybin; Demoralization; Terminal Illness; Cancer related terminal illness; psychotherapy; Terminal Cancer; Cancer Terminal
MeSH Terms: interventions — Psilocybin; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PATH (Experimental): The research study procedures include screening for eligibility, and study intervention including preparation, evaluations, one psilocybin session and follow up visits.
  -The treatment regimen consists of a single administration of psilocybin 25 mg orally combined with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions
  Interventions: Drug: Psilocybin; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Psilocybin — Oral, single administration, dosage 25 mg orally
Behavioral: Psychotherapy — The treatment regimen consists of a single administration of psilocybin orally combined with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions

SUMMARY:
The overall objective of this study is to develop and pilot test a novel regimen of psilocybin-assisted psychotherapy for demoralization in patients receiving hospice care.

-The name of the study drug involved in this study is Psilocybin

DETAILED DESCRIPTION:
The purpose of this research is to understand how psilocybin-assisted therapy may be adapted in the context of hospice care, in order to test its safety in people with terminal illness who experience demoralization, and to study how well it works to lessen symptoms of psychological and existential distress.

* This research study involves a combined drug and psychotherapeutic (talk therapy) intervention. The research study procedures include screening for eligibility, and study intervention including preparation, evaluations, one psilocybin session and follow up visits.

  * The treatment regimen consists of a single administration of psilocybin with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions
  * The name of the study drug involved in this study is Psilocybin. Psilocybin is a naturally occurring psychedelic drug produced by more than 200 species of mushrooms, which is manufactured for medical use to control potency and purity.
* Participants will be followed for up to 24 weeks (approximately 6 months) after the study treatment. It is expected that about 15 people will take part in this research study.
* This research study is a Feasibility Study, which mean it is the first time investigators are examining psilocybin-assisted therapy in the context of hospice care. Psilocybin is an "Investigational" drug, meaning that the study drug has not been approved by the U.S. Food and Drug Administration (FDA) as a treatment for any disease. However, the FDA has granted psilocybin the status of "breakthrough therapy" in the treatment of depression and the investigators have permission from the FDA to use this drug in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in hospice care at home
* Age ≥ 21 years.
* Any terminal illness with respect of exclusion criteria
* Palliative Performance Scale (PPS) ≥ 50 % (see Appendix A)
* Moderate-to-severe demoralization as measured by Demoralization Scale-II ≥ 8
* Significant other or other caregiver present at home the night of study drug administration
* No driving for 24 hours following study drug administration.
* English proficiency
* Ability to understand and the willingness to sign a written informed consent document.
* Psilocybin is very likely to have no genotoxic effects. One study that directly focused on the mutagenic potential of psilocybin did not found this type of toxicity. However, due to the lack of clinical and non-clinical studies on the effects of psilocybin on the developing human fetus, women and men of child-bearing potential and who are sexually active must agree to use an acceptable contraceptive method (hormonal or barrier method of birth control; abstinence) throughout their participation in the study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of psilocybin administration.

Exclusion Criteria:

* Current General Inpatient (GIP) hospice status
* Patients currently receiving chemotherapy
* Condition impairing oral intake or digestive absorption
* Presence of a delirium diagnosed by the CAM
* Significant suicide risk as defined by suicidal ideation with intend and a plan as endorsed on item 5 on the C-SSRS within the past month or at V0
* Current or past history of schizophrenia, psychotic disorder, bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, or borderline personality disorder, as assessed by medical history
* Patients with first-degree relatives with schizophrenia or bipolar disorder
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to psilocybin
* Other personal circumstances and behavior that would limit compliance with study requirements, or judged by the study psychiatrist and/or principal investigator to be incompatible with establishment of rapport or safe exposure to psilocybin
* Potential for adverse drug-drug interactions. Concomitant medications with significant potential to interact with study medications will be exclusionary if they cannot be tapered. These include the following:

  * Serotoninergic antidepressants
  * Centrally-acting serotonergic agents (e.g. MAO inhibitors)
  * Antipsychotics (e.g. first and second generation)
  * Mood stabilizers (e.g. lithium, valproic acid)
  * Aldehyde dehydrogenase inhibitors (e.g. disulfiram)
  * Significant inhibitors of UGT 1A0 or UGT 1A10
* Any psychiatric medication will be tapered if possible in an appropriate fashion to avoid withdrawal effects. They will be discontinued long enough before the psilocybin Session to avoid the possibility of any drug-drug interaction (the interval will be at least five times the particular drug and active metabolites' half-life).
* End stage liver disease or cirrhosis as primary hospice diagnosis
* Patients who have elevated AST and ALT five times above the normal laboratory limit on their last available bloodwork and patients with symptoms suggestive of liver failure including confusion, asterixis or jaundice.
* Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal condition or any other unstable condition that, in the opinion of the principal investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study. This may include but is not limited to clinical symptoms or recent history of significant tachyarrhythmias; severe angina or myocardial ischemia; poorly controlled congestive heart failure; poorly controlled hypertension; poorly controlled hypo- or hyperthyroidism; uncontrolled diabetes; severe renal or liver disfunction; acute respiratory failure; sepsis; history of cerebral aneurysms; glaucoma; increased intracranial pressure and any intracranial mass.
* Women who are pregnant, nursing, or planning a pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Beaussant, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Care Dimensions, Danvers, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population will include 15 adult patients, 21 years or older, who receive hospice care at home from Care Dimensions hospice in Massachusetts. The study team will screen potential participants by reviewing new admissions and reviewing the current census on a reoccurring basis. For potentially eligible patients, the study team will contact a referent hospice clinician (nurse case manager or physician) to discuss the patient case and confirm the possibility to further the consent process.
Pre-assignment Details: If the participant is being treated with psychiatric drugs at the time they are recruited, they will discuss medication tapering with the study psychiatrist and the hospice physician. If needed, the drugs will then be tapered in an appropriate fashion to avoid withdrawal effects. They will be discontinued long enough before the first Experimental Session to avoid the possibility of any drug-drug interaction (the interval will be >/= 5x the particular drug and active metabolites' half-life).
Groups:
- PATH: The research study procedures include screening for eligibility, and study intervention including preparation, evaluations, one psilocybin session and follow up visits.
  -The treatment regimen consists of a single administration of psilocybin 25 mg orally combined with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions
  Psilocybin: Oral, single administration, dosage 25 mg orally
  Psychotherapy: The treatment regimen consists of a single administration of psilocybin orally combined with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions
Period: Overall Study
Arm/Group | PATH
Started | 15
Completed | 10
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | PATH
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Relationship Status [Count of Participants; unit: Participants]
  Divorced/Separated | 2
  Married /long-term partner | 7
  Single, never married | 3
  Widowed/Loss of long-term partner | 3
Education [Count of Participants; unit: Participants]
  11th Grade or less | 1
  High school graduate or GED | 2
  2 years of college /technical school | 3
  College graduate (BS or BA) | 5
  Master's degree | 2
  Doctorate/Medical degree/Law degree | 2
Diagnosis [Count of Participants; unit: Participants]
  Gastro-intestinal cancers | 9
  Breast Cancer | 1
  GYN cancers | 1
  Light chain amyloidosis | 1
  Pulmonary fibrosis | 2
  Chronic lung allograft rejection | 1
Baseline Palliative Performance Scale [Mean (Standard Deviation); unit: units on a scale] — The Palliative Performance Scale (PPS) is a clinician-rated tool measuring functional status in palliative care. Scores range from 0% (death) to 100% (full function), in 10% increments. It assesses ambulation, activity, self-care, intake, and consciousness. Higher scores indicate better function; lower scores reflect decline. The PPS yields a single score (no subscales), based on clinical judgment. Unit of measure: scores on a scale.
  units on a scale | 62 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Screened Per Study Period
Description: This measurement will assess enrollment feasibility based on the screening log.
Time Frame: Through study completion, through 22 months
Population: Home hospice population
Measure: Number; unit: participants
Groups:
- Psilocybin- Single Arm: The research study procedures include screening for eligibility, and study intervention including preparation, evaluations, one psilocybin session and follow up visits.
  -The treatment regimen consists of a single administration of psilocybin 25 mg orally combined with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions
  Psilocybin: Oral, single administration, dosage 25 mg orally
  Psychotherapy: The treatment regimen consists of a single administration of psilocybin orally combined with a supportive psychotherapy including 2 preparation sessions and 2 integration sessions
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 4607
participants | 4607

2. Primary Outcome: Eligible Population
Description: Number of screened hospice patients who met pre-eligibility criteria and were approached for consent
Time Frame: Through study completion, over 22 months
Measure: Count of Participants; unit: Participants
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 4607
Participants | 66

3. Primary Outcome: Number of Participants Enrolled Over Study Period
Description: This measurement will assess enrollment feasibility based on the screening log.
Time Frame: Through study completion, over 22 months
Measure: Number; unit: participants
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 66
participants | 15

4. Primary Outcome: Average Time From Screening to Enrollment
Description: This measurement will assess enrollment feasibility based on the screening log.
Time Frame: From date of screening until the date of enrollment, assessed up to 12 months
Population: Participants who were enrolled in the study.
Measure: Mean (Full Range); unit: days
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 15
days | 36.6 [2 to 107]

5. Primary Outcome: Number of Therapy Sessions Completed by Enrolled Participants
Description: Therapy sessions included 5 sessions: 2 preparation visits (V1 and V2), dosing (V3) and 2 integration visits (V4 and V5)
Time Frame: Through study completion, a period of 22 months
Measure: Count of Participants; unit: Participants
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 15
Participants
  All Visits Completed | 9
  V1 through V4 completed | 1
  V1 and V2 completed | 3
  V1 completed | 1
  No therapy session completed | 1

6. Primary Outcome: Mean Score of Acceptability Ratings on Reactions to Research Participation Questionnaire Revised (RRPQR)
Description: The RRPQ-R is a validated 23-item instrument designed to assess participants' experiences and perceptions of research participation. It comprises five subscales: participation (7 items, range 7-35), personal benefit (5 items, range 5-25), emotional reactions (6 items, range 6-30), perceived drawbacks (3 items, range 3-15), and global evaluation (2 items, range 2-10). Items are rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Higher scores on participation, personal benefit, and global evaluation indicate more positive perceptions, while higher scores on emotional reactions and perceived drawbacks reflect greater negative emotional or practical impact. A total score can be calculated by summing across all items (range 23-115), with higher scores reflecting more favorable overall experiences of research participation.
Time Frame: At Week 1 post dosing session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 9
score on a scale | 90.1 (11.98)

7. Secondary Outcome: Change in Global Quality Life Score as Assessed by Functional Assessment of Chronic Illness Therapy - Palliative Care 14 (FACIT-Pal 14)
Description: The FACIT-Pal-14 is a validated 14-item measure of quality of life in palliative care populations. Items assess physical, emotional, social, and functional well-being over the past 7 days using a 5-point Likert scale (0 = not at all to 4 = very much). Scores are summed to produce a total score ranging from 0 to 56, with higher scores reflecting better quality of life. Subscale scores are not typically reported separately, but can be derived if needed by summing relevant items. The measure is widely used in palliative and supportive care research to evaluate patient-centered outcomes.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale
  Baseline | 26.5 [22.1 to 30.9]
  Week 1 (V5): number analyzed (Participants) | 9
  Week 1 (V5) | 26.9 [22.35 to 31.43]
  Week 3 (V6a): number analyzed (Participants) | 6
  Week 3 (V6a) | 30.3 [26.84 to 33.82]
  Week 7 (V6b): number analyzed (Participants) | 5
  Week 7 (V6b) | 30.8 [21.74 to 39.86]

8. Secondary Outcome: Change in Physical Domain Score as Assessed by PROMIS Pain Interference Scale (PIS)
Description: The PROMIS Pain Interference Scale (8a) is a validated 8-item instrument assessing the extent to which pain hinders engagement in social, emotional, cognitive, and physical activities. Items are rated over the past 7 days on a 5-point Likert scale (1 = not at all to 5 = very much). Raw scores range from 8 to 40 and are converted to standardized T-scores (mean = 50, SD = 10) using PROMIS scoring manuals. Higher scores indicate greater interference of pain with daily functioning. The measure is administered only if pain is reported and allows both raw and T-score interpretations to facilitate comparison across studies.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants who completed the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 9
score on a scale
  Baseline | 24.1 [17.58 to 30.64]
  Week 1 (V5): number analyzed (Participants) | 7
  Week 1 (V5) | 24.4 [15.66 to 33.2]
  Week 3 (V6a): number analyzed (Participants) | 3
  Week 3 (V6a) | 19.7 [3.13 to 36.21]
  Week 7 (V6b): number analyzed (Participants) | 4
  Week 7 (V6b) | 26.5 [11.95 to 41.05]

9. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS A and D) Score
Description: It is a self-report questionnaire consisting of 14 items, and subjects rate how they felt during the previous week on a 4-point Likert scale. The HADS consists of an anxiety and depression subscale (0-21 points each), and total scores can range from 0 to 42. Higher scores indicate more severe depression and anxiety.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants who completed the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale
  HADS-A: Baseline | 9.7 [8.01 to 11.39]
  HADS-A: Week 1 (V5): number analyzed (Participants) | 9
  HADS-A: Week 1 (V5) | 9 [5.48 to 12.52]
  HADS-A: Week 3 (V6a): number analyzed (Participants) | 6
  HADS-A: Week 3 (V6a) | 5.67 [1.13 to 10.2]
  HADS-A: Week 7 (V6b): number analyzed (Participants) | 5
  HADS-A: Week 7 (V6b) | 8 [4.28 to 11.72]
  HADS-D: Baseline | 10.1 [7.54 to 12.66]
  HADS-D: Week 1 (V5): number analyzed (Participants) | 9
  HADS-D: Week 1 (V5) | 9.67 [6.41 to 12.93]
  HADS-D: Week 3 (V6a): number analyzed (Participants) | 6
  HADS-D: Week 3 (V6a) | 7.83 [3.88 to 11.78]
  HADS-D: Week 7 (V6b): number analyzed (Participants) | 5
  HADS-D: Week 7 (V6b) | 8.2 [2.83 to 13.57]

10. Secondary Outcome: Change in Life Attitude Profile - Revised, Death Acceptance Subscale (LAP-R) Score
Description: The LAP-R Death Acceptance subscale is a validated 8-item measure assessing acceptance of and anxiety about death. Items are rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). Subscale scores are calculated by summing item responses, yielding a total range of 9 to 56, with higher scores reflecting greater acceptance of death and lower death-related anxiety. The measure is commonly used in palliative care and existential research to evaluate psycho-existential adjustment in serious illness.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants who completed the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 9
score on a scale
  Baseline | 32.3 [24.83 to 39.85]
  Week 1 (V5): number analyzed (Participants) | 1
  Week 1 (V5) | 35
  Week 3 (V6a): number analyzed (Participants) | 4
  Week 3 (V6a) | 34.5 [14.77 to 54.23]
  Week 7 (V6b): number analyzed (Participants) | 0

11. Secondary Outcome: Challenging Experience Questionnaire (CEQ) Score
Description: The CEQ is a validated 26-item instrument assessing psychologically and somatically difficult aspects of psilocybin experiences. It consists of seven subscales: grief (3 items, range 3-15), fear (6 items, range 6-30), death (3 items, range 3-15), insanity (3 items, range 3-15), isolation (3 items, range 3-15), physical distress (3 items, range 3-15), and paranoia (5 items, range 5-25). Items are rated on a 5-point Likert scale (1 = not at all to 5 = extremely). Subscale scores are computed by summing responses within each domain, with higher scores indicating more challenging experiences. A total score (range 26-130) may also be calculated by summing across all items, providing a global index of psychological challenge.
Time Frame: Immediately after the intervention, at the end of the dosing day
Population: Treated participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale | 36.6 (20.8)

12. Secondary Outcome: Change in Social Isolation Scale (SIS) Score
Description: The PROMIS Social Isolation Scale-6a is a validated 6-item short form that measures perceived social disconnection, including feelings of exclusion, detachment, and lack of belonging. Items are rated on a 5-point Likert scale (1 = never to 5 = always). Raw scores range from 6 to 30 and are converted to standardized T-scores (mean = 50, SD = 10) based on PROMIS scoring guidelines. Higher scores represent greater perceived social isolation. The measure is widely used in psychosocial and palliative care research to assess the impact of illness on social well-being.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants who completed the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale
  Baseline | 14.9 [12.15 to 17.65]
  Week 1 (V5): number analyzed (Participants) | 9
  Week 1 (V5) | 15.6 [12.05 to 19.06]
  Week 3 (V6a): number analyzed (Participants) | 6
  Week 3 (V6a) | 13.5 [8.96 to 18.04]
  Week 7 (V6b): number analyzed (Participants) | 5
  Week 7 (V6b) | 13.4 [8.54 to 18.26]

13. Secondary Outcome: Change in Spiritual Domain Score as Assessed by Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being 12 (FACIT-sp-12)
Description: The FACIT-Sp-12 is a validated 12-item measure widely used in cancer and palliative care to assess spiritual well-being. It includes three subscales: meaning (4 items, range 0-16), peace (4 items, range 0-16), and faith (4 items, range 0-16). Items are rated on a 5-point Likert scale (0 = not at all to 4 = very much). Subscale scores are summed, and a total score (range 0-48) is obtained by summing across all items. Higher scores indicate greater spiritual well-being. The FACIT-Sp-12 is one of the most commonly used measures of spirituality in serious illness research and has strong psychometric validity.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants who completed the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale
  Baseline | 22.3 [17.51 to 27.09]
  Week 1 (V5): number analyzed (Participants) | 9
  Week 1 (V5) | 26.7 [21.81 to 31.53]
  Week 3 (V6a): number analyzed (Participants) | 6
  Week 3 (V6a) | 30.3 [20.84 to 39.83]
  Week 7 (V6b): number analyzed (Participants) | 5
  Week 7 (V6b) | 29.4 [18.63 to 40.17]

14. Secondary Outcome: Change in Demoralization Scale (DS-II)
Description: The DS-II is a validated 16-item self-report measure of demoralization, capturing experiences of disheartenment, helplessness, and loss of meaning. It comprises two subscales: meaning and purpose (8 items, range 0-16) and distress and coping ability (8 items, range 0-16). Items are rated on a 3-point scale (0 = never, 1 = sometimes, 2 = often). Subscale scores are summed, and a total score (range 0-32) is calculated by adding across all items, with higher scores indicating greater demoralization. For Version 5 (V5), items are anchored to the past week rather than the past two weeks in the original version, improving temporal sensitivity in clinical research.
Time Frame: At Baseline, and weeks 1, 3, and 7
Population: Treated participants who completed the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale
  Baseline | 17.3 [13.17 to 21.43]
  Week 1 (V5): number analyzed (Participants) | 9
  Week 1 (V5) | 12 [7.02 to 16.98]
  Week 3 (V6a): number analyzed (Participants) | 6
  Week 3 (V6a) | 8.5 [2.25 to 14.75]
  Week 7 (V6b): number analyzed (Participants) | 5
  Week 7 (V6b) | 14.6 [2.07 to 27.13]

15. Secondary Outcome: Mystical Experience Questionnaire (MEQ-30)
Description: The MEQ-30 is a validated 30-item self-report instrument assessing the phenomenological features of mystical-type experiences induced by psychedelics. It yields four subscales: mystical (15 items, range 0-75), positive mood (6 items, range 0-30), transcendence of time and space (6 items, range 0-30), and ineffability (3 items, range 0-15). Items are rated on a 6-point Likert scale (0 = none to 5 = extreme). Subscale scores are summed, and a total score (range 0-150) is calculated by summing across all items. Higher scores indicate stronger mystical-type experiences, with ≥60% of the maximum possible score on each subscale often used as a criterion for a "complete" mystical experience.
Time Frame: Immediately after the intervention, at the end of the dosing day
Population: Treated participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin- Single Arm
Number analyzed (Participants) | 10
score on a scale | 84.1 (34.47)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Psilocybin- Single Arm
All-Cause Mortality (participants affected / at risk) | 9/15
Serious Adverse Events (participants affected / at risk) | 10/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin- Single Arm (N=15)
Ascites (Gastrointestinal disorders) | 1 (1) — First episode of symptomatic ascites (pain, nausea, vomiting and shortness of breath) leading to admission at hospice facility as GIP during one week. Related to terminal illness (bile duct cancer).
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Increased Abdominal Pain related to terminal illness progression (colon cancer with mets to liver and lung) - Admitted GIP at the Hospice House for complex pain management. Patient was Off Treatment at that time.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Sudden episode of dyspnea around 5pm, resulting in death shortly after.
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant fell at his home and fractured his right femoral neck. Hospitalization required.
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Progressive decline due to underlying disease (lung fibrosis). Patient found to be deceased by son on morning of 1/8/23. At this time, patient was Off Treatment after completing the therapeutic intervention per protocol.
Cardiac arrest (Cardiac disorders) | 5 (5) — Death occured due to terminal illness progression.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Increased dyspnea, somnolence and confusion at home despite O2 5L. GIP admission for end of life symptom management. Participant passed away due to terminal illness progression (interstitial lung disease).
Depressed level of consciousness (Nervous system disorders) | 1 (1) — Patients found unconscious on the floor.
Pain (General disorders) | 1 (1) — Significant increase of pain necessiting GIP admission.
Nausea (Gastrointestinal disorders) | 1 (1) — Nausea. At this time, patient was Off Treatment after completing the therapeutic intervention per protocol.
Fatigue (General disorders) | 1 (1) — Noted weakness in patient chart. At this time, patient was Off Treatment after completing the therapeutic intervention per protocol.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin- Single Arm (N=15)
Fatigue (General disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (5)
Hypoglycemia (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9)
Sedation (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Anger (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Crying (Psychiatric disorders) | 7 (7)
Depression (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This pilot study is limited by its small sample size, lack of control group, and homogeneous participant demographics. Its single-site design further limits generalizability. Additionally, due to the rapidly evolving clinical condition of participants, missing data at later time points limited our ability to assess medium to long-term outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04950608/Prot_SAP_000.pdf